CLINICAL TRIAL: NCT03819894
Title: Hs-cTn - Optimizing the Diagnosis of Acute Myocardial Infarction/Injury in Women
Acronym: CODE-MI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BC Centre for Improved Cardiovascular Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: H18-02116
Record Dates: First submitted 2019-01-21; First posted 2019-01-29 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarction; Sex Differences; High Sensitivity Troponin
Keywords: myocardial infarction; sex differences; high-sensitivity cardiac troponin; biomarkers; heart attack; emergency department; acute coronary syndrome
MeSH Terms: conditions — Myocardial Infarction; Emergencies; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized trial. Unidirectional crossover design where clusters cross over sequentially, in random order, from the control to intervention phase.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is the introduction of a lower female threshold. In cluster-randomized trials, the cluster (i.e., hospital) is the unit of randomization.
  Interventions: Diagnostic Test: Introduction of a lower female hs-cTn threshold
- Control (No Intervention): The control phase will be standard of care, with the use of an overall population hs-cTn T and I threshold, for both men and women, to identify those with myocardial injury/infarction.

INTERVENTIONS:
Diagnostic Test: Introduction of a lower female hs-cTn threshold — The new female hs-cTn threshold will be baed on current recommendations for each of the assays used (hs-cTn T and I). The hospitals are the unit of randomization. At 5-month intervals, randomly selected hospitals will be advised that they are to transition to the intervention phase. For all men, the standard of care, overall population threshold will be used throughout the entire study.
  Arms: Intervention

SUMMARY:
The project is focussed on evaluating the impact of using a female-specific threshold in the diagnosis of myocardial infarction. This female threshold is lower than the overall hs-cTn threshold currently in use. The investigators hypothesize that this change in process, applied at the hospital level, will lead to better assessment, treatment and outcomes of women presenting to the emergency department with chest pain that is cardiac in nature.

DETAILED DESCRIPTION:
In subjects with suspected acute coronary syndromes (ACS), females are significantly less likely to undergo investigations, receive evidence-based treatments, and consistently have worse outcomes than males. The gap in outcomes is particularly marked among adults < 55 years of age. Sex differences in symptom presentation and in the diagnostic threshold for cardiac biomarkers have been suggested as reasons for the under-diagnosis and under-treatment of women. Cardiac troponin (cTn) T and I are proteins specific to the myocardium, which with elevated and changing concentrations detected in the blood, along with signs or symptoms consistent with myocardial ischemia, are indicative of a diagnosis of myocardial infarction (MI). With the introduction of high-sensitivity (hs) cTn tests, which allow the detection of very low concentrations of troponin, it has become evident that the level of cTn in a healthy population is approximately two-fold higher in males than in females.

Consequently, the 99th percentile threshold for cTn, the reference value used in diagnosis of MI, is lower in females compared to males. Despite this evidence and recent guidelines recommending the use of sex specific thresholds, a single, overall cTn threshold is still being used for diagnosis of MI, in both men and women, in most clinical settings.

There is mounting evidence from several jurisdictions that the rate of MI is increasing among younger females, and that there is a persistent under-diagnosis, under-treatment, and high risk of adverse outcomes among females, especially younger females, compared to their male counterparts. A better approach to the diagnostic assessment of females presenting to the emergency department (ED) with chest pain is therefore urgently needed. Additionally, several Canadian hospitals have recently made the transition from sensitive to high sensitivity cTn assays, allowing for the examination of subtle but important sex-specific differences in cTn concentrations. With this background, the investigators propose a nationwide, randomized clinical trial (RCT) to determine whether establishing female thresholds results in improved diagnosis and treatment of MI and therefore improved prognosis in women.

To determine whether the use of female hs-cTn thresholds in the assessment of women presenting to the ED with chest pain suggestive of cardiac ischemia, improves diagnostic assessment, treatment and 2-year outcomes. Specifically, the investigators will examine the impact of using female hs-cTn thresholds on:

* Diagnostic and therapeutic strategies;
* Prognosis: 2-year all-cause mortality, non-fatal MI, incident heart failure (HF) hospitalization or emergent/urgent coronary revascularization;
* Costs of diagnostic testing and treatment.

ELIGIBILITY:
Inclusion Criteria:

* >20 years of age
* Present to the ED with chest pain or shortness of breath suggestive of ischemia
* Have a valid personal health identifier
* Have 1 hs-cTn test result

Exclusion Criteria:

* Have ST elevation myocardial infarction (STEMI)
* Not residents in the same province as the hospital ED to which they present or move out of province within a year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24000 (Estimated)
Dates: Start 2020-02-08 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with all-cause mortality, non-fatal myocardial infarction, hospitalization for incident heart failure, or urgent/emergent coronary revascularization (percutaneous coronary intervention or coronary artery bypass surgery) | 2-year post index emergency department presentation
  Composite of all-cause mortality, re-admission for non-fatal MI, incident HF, or urgent/emergent coronary revascularization

SECONDARY OUTCOMES:
Number of patients with a) Non-fatal myocardial infarction or all-cause mortality; b) Urgent/emergent coronary revascularization or all-cause mortality; c) Hospitalization for heart failure or all-cause mortality. | 2-year post index emergency department presentation
  The secondary outcomes include the individual components of the composite outcome with death, to account for competing risk.
Proportion of patients who fill at least one prescription for evidence-based cardiac medications | Within 90 days of ED visit
  Medications include beta-blockers, Angiotensin Converting Enzyme (ACE)-I/Angiotensin II receptor blockers (ARB), statins, anti-platelets
Proportion of patients who undergo diagnostic tests | Within 90 days of ED visit
  Diagnostic tests include nuclear medicine cardiac scan, exercise stress test, diagnostic cardiac catheterization/CT angiogram or echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Karin Humphries, DSc, Principal Investigator — Medicine, Cardiology, UBC, BC Centre for Improved Cardiovascular Health
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Zhao Y, Izadnegahdar M, Lee MK, Kavsak PA, Singer J, Scheuermeyer F, Udell JA, Robinson S, Norris CM, Lyon AW, Pilote L, Cox J, Hassan A, Rychtera A, Johnson D, Mills NL, Christenson J, Humphries KH. High-Sensitivity Cardiac Troponin-Optimizing the Diagnosis of Acute Myocardial Infarction/Injury in Women (CODE-MI): Rationale and design for a multicenter, stepped-wedge, cluster-randomized trial. Am Heart J. 2020 Nov;229:18-28. doi: 10.1016/j.ahj.2020.06.013. Epub 2020 Jun 25. PMID 32916606